CLINICAL TRIAL: NCT02848677
Title: Serum Levels of Advanced Glycation End-products After Dietary Intervention in Hypertensive Patients: Study Protocol of a Randomized Clinical Trial.
Brief Title: Serum Levels of Advanced Glycation End-products After Dietary Intervention in Hypertensive Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 150325
Record Dates: First submitted 2016-07-26; First posted 2016-07-28 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Hypertension,
Keywords: advanced glycation end-products; Cardiovascular disease; Low Sodium Diet; vascular inflammation
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention group (Active Comparator): Nutritional counseling implemented by a dietitian for a low sodium diet rich in fruits, vegetables, low fat dairy foods, and low in processed foods.
  Interventions: Behavioral: Nutritional counseling
- control group (Sham Comparator): usual care of hypertensive patients.
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: Nutritional counseling — Nutritional counseling implemented by a dietitian for a low sodium diet rich in fruits, vegetables, low fat dairy foods, and low in processed foods.
  Arms: intervention group
Behavioral: usual care — usual care of hypertensive patients.
  Arms: control group

SUMMARY:
Cardiovascular disease (CVD) is considered the main cause of mortality in the western world. There are many factors that contribute to the onset and progression of cardiovascular disease, including hypertension. Hypertension is a multi-factorial condition that includes nutritional disorders in its causality line. It is believed that advanced glycation end-products (AGEs) is one of the pathophysiological causes that explain the occurrence of high blood pressure in diabetic patients. This study has the role of describing the protocol of a randomized clinical trial aiming to evaluate changes in serum levels of end products of advanced glycation after an intervention for eating habit changes in hypertensive individuals.

The investigators designed a randomized clinical trial, with non-blinded assessment of outcomes. Participants will be recruited from the outpatient clinic for hypertension of a public hospital in Porto Alegre, aged from 40 to 80 years old and without diabetes. Hypertension is defined as systolic blood pressure ≥ 140 mmHg, diastolic blood pressure ≥ 90 mmHg, or antihypertensive medication use. Participants will be assigned to one of two groups. The intervention group will receive monthly educational intervention sessions for low salt diet, high in fruits and vegetables, and low in processed foods for a period of 6 months. Besides these, the intervention group will receive a standard telephone interview every two weeks to motivate them to follow the diet. The control group will receive the usual counseling for low sodium diet in monthly appointment with a dietitian, following the hypertension care clinic protocol.

This study aims to investigate if there are significant changes in serum levels of advanced glycation end products, after the nutritional intervention with diet guidance in fruits, vegetables, low in sodium and processed foods in hypertensive patients because several studies have shown that less processed food rich in antioxidants with low sodium content, play an important role in reducing levels of AGEs which are precursors of vascular inflammation and progression of cardiovascular diseases.

DETAILED DESCRIPTION:
There will be a randomized, non-blinded, parallel-group clinical trial comparing serum AGESs level in patients randomized to receive an educational program of diet counseling or the usual care.

Study population: Hypertensive patients attending the outpatient clinic for hypertension treatment at a university-affiliated hospital in southern Brazil.

Intervention group - Nutritional counseling implemented by a dietitian for a low sodium diet rich in fruits, vegetables, low fat dairy foods, and low in processed foods. Patients will be evaluated every month.

Control group - usual care of hypertensive patients. Patients will be evaluated after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* It will be included patients aged between 40 and 80 years old,
* diagnosed with hypertension defined by systolic blood pressure ≥ 140 mmHg, diastolic blood pressure ≥ 90 mmHg,
* or the use of drugs for hypertension; patients not following nutritional counseling in the last 6 months.

Exclusion Criteria:

* will be patients with inflammatory diseases, receiving chemotherapy treatment,
* diagnosed with diabetes mellitus,
* referred for nutritional counseling or unable to conduct the interview and to participate in the intervention program,
* pregnant women and nursing mothers.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-11 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
reduction of serum levels of AGEs | 6 months

SECONDARY OUTCOMES:
Changes from baseline and six months in blood pressure | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Leila B Moreira, MD PHD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Leila Beltrami Moreira, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Prasad C, Imrhan V, Marotta F, Juma S, Vijayagopal P. Lifestyle and Advanced Glycation End Products (AGEs) Burden: Its Relevance to Healthy Aging. Aging Dis. 2014 Jun 1;5(3):212-7. doi: 10.14336/AD.2014.0500212. eCollection 2014 Jun. PMID 24900944
- [Result] Ward MS, Fortheringham AK, Cooper ME, Forbes JM. Targeting advanced glycation endproducts and mitochondrial dysfunction in cardiovascular disease. Curr Opin Pharmacol. 2013 Aug;13(4):654-61. doi: 10.1016/j.coph.2013.06.009. Epub 2013 Jul 16. PMID 23871446
- [Result] Gul A, Rahman MA, Salim A, Simjee SU. Advanced glycation end-products in senile diabetic and non-diabetic patients with cardiovascular complications. Age (Dordr). 2008 Dec;30(4):303-9. doi: 10.1007/s11357-008-9072-1. Epub 2008 Sep 3. PMID 19424854
- [Result] Erdine S, Ari O, Zanchetti A, Cifkova R, Fagard R, Kjeldsen S, Mancia G, Poulter N, Rahn KH, Rodicio JL, Ruilope LM, Staessen J, van Zwieten P, Waeber B, Williams B. ESH-ESC guidelines for the management of hypertension. Herz. 2006 Jun;31(4):331-8. doi: 10.1007/s00059-006-2829-3. PMID 16810473
- [Result] Nobre F. [Introduction: Brazilian guidelines on hypertension VI. Brazilian Society of Cardiology, Brazilian Society of Hypertension, Brazilian Society of Nephrology]. J Bras Nefrol. 2010 Sep;32 Suppl 1:III. doi: 10.1590/s0101-28002010000500002. No abstract available. Portuguese. PMID 22262215
- [Result] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; National Heart, Lung, and Blood Institute Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure; National High Blood Pressure Education Program Coordinating Committee. The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure: the JNC 7 report. JAMA. 2003 May 21;289(19):2560-72. doi: 10.1001/jama.289.19.2560. Epub 2003 May 14. PMID 12748199
- [Result] Lewington S, Clarke R, Qizilbash N, Peto R, Collins R; Prospective Studies Collaboration. Age-specific relevance of usual blood pressure to vascular mortality: a meta-analysis of individual data for one million adults in 61 prospective studies. Lancet. 2002 Dec 14;360(9349):1903-13. doi: 10.1016/s0140-6736(02)11911-8. PMID 12493255
- [Result] Vasdev S, Stuckless J, Richardson V. Role of the immune system in hypertension: modulation by dietary antioxidants. Int J Angiol. 2011 Dec;20(4):189-212. doi: 10.1055/s-0031-1288941. PMID 23204821
- [Result] Bodiga VL, Eda SR, Bodiga S. Advanced glycation end products: role in pathology of diabetic cardiomyopathy. Heart Fail Rev. 2014 Jan;19(1):49-63. doi: 10.1007/s10741-013-9374-y. PMID 23404649
- [Result] Dhar I, Dhar A, Wu L, Desai KM. Methylglyoxal, a reactive glucose metabolite, increases renin angiotensin aldosterone and blood pressure in male Sprague-Dawley rats. Am J Hypertens. 2014 Mar;27(3):308-16. doi: 10.1093/ajh/hpt281. Epub 2014 Jan 16. PMID 24436324
- [Result] Finot PA. Historical perspective of the Maillard reaction in food science. Ann N Y Acad Sci. 2005 Jun;1043:1-8. doi: 10.1196/annals.1333.001. PMID 16037216
- [Result] Kwak EJ, Lim SI. The effect of sugar, amino acid, metal ion, and NaCl on model Maillard reaction under pH control. Amino Acids. 2004 Aug;27(1):85-90. doi: 10.1007/s00726-004-0067-7. Epub 2004 Feb 27. PMID 15309575
- [Result] Poulsen MW, Bak MJ, Andersen JM, Monosik R, Giraudi-Futin AC, Holst JJ, Nielsen J, Lauritzen L, Larsen LH, Bugel S, Dragsted LO. Effect of dietary advanced glycation end products on postprandial appetite, inflammation, and endothelial activation in healthy overweight individuals. Eur J Nutr. 2014;53(2):661-72. doi: 10.1007/s00394-013-0574-y. Epub 2013 Aug 9. PMID 23929260
- [Result] d'Almeida KS, Souza GC, Rabelo-Silva ER. Validity and reliability of the Dietary Sodium Restriction Questionnaire (DSRQ). Nutr Hosp. 2013 Sep-Oct;28(5):1702-9. doi: 10.3305/nh.2013.28.5.6679. PMID 24160236
- [Result] Wu ET, Liang JT, Wu MS, Chang KC. Pyridoxamine prevents age-related aortic stiffening and vascular resistance in association with reduced collagen glycation. Exp Gerontol. 2011 Jun;46(6):482-8. doi: 10.1016/j.exger.2011.02.001. Epub 2011 Feb 18. PMID 21316441
- [Result] Barbosa JH, Oliveira SL, Seara LT. [The role of advanced glycation end-products (AGEs) in the development of vascular diabetic complications]. Arq Bras Endocrinol Metabol. 2008 Aug;52(6):940-50. doi: 10.1590/s0004-27302008000600005. Portuguese. PMID 18820805